CLINICAL TRIAL: NCT07099794
Title: Liposomal Irinotecan (II) and Fluorouracil and Calcium Folinate in Combination With or Without Renvastinib for Second-line Treatment of Advanced Biliary System Tumors: a Randomized, Two-cohort, Prospective Phase II Study
Brief Title: A Randomized, Two-cohort, Prospective Phase II Clinical Study of the Second-line Treatment of Advanced Biliary System Tumors With Liposomal Irinotecan (II) Combination Regimen
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC EC/IRB
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-06

CONDITIONS: Biliary Tract Cancer (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NALIRI+Lenvatinib (Experimental): Liposomal irinotecan+5-FU/LV+Lenvatinib
  Interventions: Drug: Liposomal irinotecan+5-FU/LV+Lenvatinib
- NALIRI (Experimental): Liposomal irinotecan+5-FU/LV
  Interventions: Drug: NALIRI

INTERVENTIONS:
Drug: Liposomal irinotecan+5-FU/LV+Lenvatinib — Liposomal irinotecan II: calculated as free base, 56.5 mg/m2, IV, d1q2w Renvastinib: ≥60kg, 12mg; <60kg, 8mg, PO, once daily 5-FU: 1200 mg/ (m2·d) x2d continuous intravenous infusion for 46-48h, q2w LV: 400 mg/m2 intravenously, d1 q2w
  Arms: NALIRI+Lenvatinib
Drug: NALIRI — Liposomal irinotecan II: calculated as free base, 56.5 mg/m2, IV, d1q2w 5-FU: 1200 mg/ (m2·d) x2d continuous intravenous infusion for 46-48h, q2w LV: 400 mg/m2 intravenously, d1 q2w
  Arms: NALIRI

SUMMARY:
This is a randomized, two-cohort, multicenter Phase II clinical study. To evaluate the efficacy and safety of liposomal irinotecan II and 5-FU/LV combined with or without renvastinib in the treatment of patients with advanced biliary system tumors, 90 patients were scheduled to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* The patients voluntarily joined the study and signed the informed consent;
* Histologically or cell line confirmed advanced biliary system malignancies, including intrahepatic, extrahepatic, and gallbladder cancers;
* Previous first-line combination therapy failed;
* At least one measurable lesion meets the RECIST v1.1 criteria
* ECOG PS：0~1；
* Expected survival ≥12 weeks;
* Essential organ and hematological function;
* Patients need contraception;

Exclusion Criteria:

* The patient had previously received irinotecan, 5-Fu, and antiangiogenic agents;
* Patients had active malignancies other than BTC within 5 years or at the same time.
* Clinical symptoms or diseases of the heart that are not well controlled;
* Patients with hypertension who cannot be reduced to the normal range by antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
* Any clinically significant gastrointestinal disorder, including bleeding, inflammation, occlusion, or diarrhea > grade 2;
* A thrombotic or embolic event occurred within 6 months prior to the start of the study therapy;
* Use of strong CYP3A4/CYP2C19 inducers including rifampicin (and its analogiaries) and hypericum perforatum or strong CYP3A4/CYP2C19 inhibitors and/or strong UGT1A inhibitors within 14 days prior to signing the informed consent;
* Known allergy to the study drug;
* An uncontrolled infection occurs during screening;
* Patients with congenital or acquired immune deficiency (e.g., HIV);
* Have a history of brain metastases or have developed brain metastases;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5 years
  The time between participant randomization and first recorded disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Patients were randomized to the time of death from any cause.
Objective Response Rate | 5 years
  The proportion of participants in the analyzed population with confirmed complete (CR) or partial response (PR) based on RECIST v1.1
Disease control rate | 5 years
  Percentage of cases with confirmed complete response, partial response, and stable disease (≥ 8 weeks) in patients for whom response could be evaluated.
Adverse events | 5 years
  Adverse events (AE)/Serious Adverse Events (SAE) (as determined by NCI-CTCAE 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No